CLINICAL TRIAL: NCT03105531
Title: Screening for Primary Aldosteronism in a Population of Patients With Hypertension
Acronym: PRIMAL
Status: Completed | Type: Observational
Sponsor: Uppsala University (Other)
Collaborators: Uppsala-Örebro Regional Research Council (Other)
Responsible Party: Principal Investigator, Per Hellman, Professor, Head of the Department of Surgical Sciences, Uppsala University, Uppsala University
Other Study IDs: Project 16-25
Record Dates: First submitted 2017-03-27; First posted 2017-04-10 (Actual); Last update posted 2023-12-04 (Actual); Status verified 2023-12

CONDITIONS: Primary Aldosteronism; Hypertension; Hypertension Secondary
Keywords: primary aldosteronism; hypertension; screening; secondary hypertension
MeSH Terms: conditions — Hyperaldosteronism; Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples from patients with documented primary aldosteronism are going to be (with the patients informed consent) obtained to be stored in Uppsala Biobank for future scientific purposes.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Primary aldosteronism (PA) is an under-diagnosed cause of arterial hypertension. Cardiovascular morbidity and mortality in hypertension rises significantly for patients who have aldosterone overproduction when compared with those with primary hypertension and the same level of blod pressure elevation. The classical signs of PA such as severe hypertension and hypokalemia may be absent, why screening in defined risk groups has been recommended. Screening has not been systematically implemented in Sweden, probably due to expensive, time and effort-consuming clinical routine protocols and low awareness of the problem among clinicians. The prevalence of PA in patients with hypertension in Sweden has not been studied adequately, and few studies from Northern Europe have addressed the problem.

The primary objective is to investigate prevalence of PA among patients with hypertension in primary care and to implement and assess optimal treatment. Discovered cases of PA will go through routine clinical work-up in order to distinguish the subtype of PA, which includes computed tomography of adrenals and adrenal vein sampling (AVS) in those willing and fit for surgical treatment. Treatment will be then chosen depending on the PA subtype. Those with unilateral disease who are willing and fit for surgery will be offered unilateral minimally invasive adrenalectomy. Patients who oppose or have contraindications to operative treatment, as well as patients with bilateral disease will be offered medical treatment with mineralocorticoid receptor antagonists (MRA).

Study participants will be then followed up one year after surgery or initiation of specific medical treatment. Please se outcome measures for relevant description of those.

Blood samples will be collected from patients with confirmed PA to be stored in a biobank for potential future genetical and biochemical studies. A subgroup of patients with PA will undergo adrenal-specific positron-emission tomography to assess the possibility to un-invasively diagnose and subtype PA.

DETAILED DESCRIPTION:
Primary care hypertensive patients corresponding to eligibility criteria will be contacted by letter (including informed consent form) and thus invited to take part in the present study. On the one hand, the letter will be sent to a group of hypertensive patients who could be identified from the hypertension diagnosis based search through the database belonging to the computerized patient journal system. On the other hand, the letter will be offered to consecutive hypertension patients who contact their primary care facility for whatever reason. The first 1200 patients who have given informed consent to participation are going to be enrolled in the study.

The study will be conducted mostly in Karlstad, a town in central Sweden with population of about 89000 people. Some of approximately 4000 hypertensive patients enlisted at one of the major primary care facilities in town, Gripen Outpatient Clinic, will be contacted in the above manner. Gripen serves totally about 21000 outpatients. If needed for enrollment purposes, one other of the regions major outpatient clinics will be involved. Aldosterone - Renin Ratio (ARR), intravenous sodium chloride (i.v. NaCl) suppression test and adrenal computed tomography (CT) will de done at Karlstad Central Hospital - at Surgical, Endocrinological and X-ray Departments, respectively. AVS is planned to be carried out at an X-ray laboratory at Uppsala University Hospital. Adrenalectomies will be performed at Surgical departments in both Uppsala and Karlstad.

After a two week run-in period with liberal salt intake and abstinence form licorice and chewing tobacco, blood samples will be taken from study participants. Sampling will be performed at 8-10 a.m., ideally 2 hrs after awakening and after 5-15 min of seated rest.

Plasma aldosterone, plasma renin (Direct Renin Concentration, DRC), serum sodium, potassium and creatinine are going to be analysed. Aldosterone-Renin Ratio (ARR) > = 50 pmol/mU and plasma aldosterone > = 170 pmol/l are the criteria that will prompt further work-up upon suspicion of PA. Patients with other test results will be considered to not have PA - if they are normokalemic and not using mineralocorticoid receptor antagonists (MRA).

Patients using MRA will be offered optimization and retest. MRA will be then discontinued for at least 6 weeks and substituted if needed with alfa- or calcium blockers. Hypokalemic patients with test results not prompting suspicion of PA will also be optimized with potassium supplementation until normokalemia is sustained before retesting.

Those with suspicion-raising ARR and aldosterone will go further in evaluation unrelated to potassium level, but will need to correct any hypokalemia prior to i.v. NaCl suppression test. Patients with suspicion of PA who have uncontrolled hypertension (with systolic blood pressure > 180 or diastolic pressure > 110 mm Hg) will need more efficient treatment before proceeding to confirmation work-up. Patients with chronic heart failure NYHA (New York Heart Association) stage > 2 are going to be excluded from i.v. NaCl suppression testing.

Possibility of PA in patients excluded from the study prior to confirmation work-up can be assessed by the criteria that may be present at the time of ARR-evaluation. Diagnosis of PA can be stated if initial hypokalemia, plasma renin below detection limit and plasma aldosterone above 550 pmol/l are encountered.

Patients with suspected PA will be offered intravenous sodium chloride (NaCl) suppression test to confirm or exclude the diagnosis.The criteria used here correspond to the criteria recommended by the last edition of An Endocrine Society Clinical Practice Guideline for management of primary aldosteronism (2016).

Intravenous sodium chloride suppression test involves intravenous administration of 2 liters of NaCl 0,9% solution given over 4 hours under medical observation. Post-test plasma aldosterone > 280 pmol/l confirms PA, aldosterone < 140 pmol/l excludes PA in normokalemic subjects. According to protocol amendment from February 2, 2018, patients with aldosterone within 140 - 280 pmol/l are going to be offered optimization with discontinuation of eventual potassium wasting diuretics, Amiloride and all other antihypertensive medication which can influence the screening test for minimum of 4 weeks besides other measures above mentioned as optimization before ARR - if those had not been effectively implemented before. After this optimization period the i.v. NaCl suppression test will be repeated. If aldosterone after this second NaCl suppression test is < 190 pmol/l, those patients will be considered free of PA and excluded form further analysis. Patients with aldosterone > = 190 pmol/l will be considered to have PA.

The patients where PA has been confirmed will be evaluated onwards as previously described.

Patients with bilateral disease will be offered medical treatment with MRA. Patients with unilateral disease (if fit and willing) will be recommended minimally invasive surgical treatment.

Treatment results are going to be followed up after one year, as detailed in the outcome measures.

ELIGIBILITY:
Inclusion Criteria:

* participants must have Swedish personal number (that gives right to all kinds of necessary planned health care)

Exclusion Criteria:

* pregnancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: An unselected population of primary care patients with hypertension
Sampling Method: Non-Probability Sample
Enrollment: 1183 (Actual)
Dates: Start 2017-04-07 (Actual); Primary Completion 2023-11-28 (Actual); Study Completion 2023-11-28 (Actual)

PRIMARY OUTCOMES:
Prevalence estimates of primary aldosteronism (PA) and of PA subtypes in a Swedish population of primary care patients with arterial hypertension | For each patient, the time necessary to go through initial (sometimes repeated) screening with ARR, then (sometimes repeated) confirmation testing with i.v. NaCl-suppression test will be approximately 6 months
  ARR - Aldosterone-Renin Ratio; i.v. - intravenous; NaCl - sodium chloride;

SECONDARY OUTCOMES:
The proportion of screening-discovered patients with PA who could be offered surgical treatment - and who have accepted operation and have been unilaterally adrenalectomized. | Considering work-up time and waiting time for planned surgery of this type it is realistic to assume minimal time frame of approximately 2 years
  Percentage - relevant to the number of discovered cases of PA.
Changes in clinical characteristics of hypertension and in antihypertensive treatment regimen still needed - one year after the diagnosis of primary aldosteronism had been stated and specific treatment applied. | Evaluation of treatment effects is done at the follow-up patient contact one year after adrenal surgery or initiation of specific medical treatment - approximately 1,5 - 2 years after the first screening.
  Those patients who get the diagnosis of PA after the initial screening and further investigations by the study protocol will be offered specific medical or surgical treatment - depending on the subtype of PA.
  In both medically and surgically treated patients the assessment is going to include blood pressure level, usage of MRA and their doses, usage of other antihypertensive medications, their number and doses, frequency of significant side effects of MRA such as gynecomastia, gynecodynia, erectile dysfunction, decreased libido, menstrual disturbances.
Serum potassium level - one year after the diagnosis of primary aldosteronism had been stated and specific treatment applied. | Evaluation is done at the follow-up patient contact one year after adrenal surgery or initiation of specific medical treatment - approximately 1,5 - 2 years after the first screening.
  Serum potassium in mmol/l.
Any potassium supplementation if still needed - one year after the diagnosis of primary aldosteronism. | Evaluation is done at the follow-up patient contact one year after adrenal surgery or initiation of specific medical treatment - approximately 1,5 - 2 years after the first screening.
  Supplementation measured as "still needed" or "not needed".
Serum creatinine - one year after the diagnosis of primary aldosteronism. | Evaluation is done at the follow-up patient contact one year after adrenal surgery or initiation of specific medical treatment - approximately 1,5 - 2 years after the first screening.
  Serum creatinine in mcmol/l.
Control of Aldosterone Renin Ratio (ARR) after the same 2 weeks long preliminary optimization period as at initial ARR screening - one year after surgical treatment for PA. | Evaluation is done at the follow-up patient contact one year after adrenal surgery - approximately 2 years after the first screening.
  As plasma aldosterone is measured in pmol/l and plasma Direct Renin Concentration (DRC) in mU/l, ARR is accordingly measured as pmol/mU. The measure of ARR will be evaluated as at the initial ARR screening.
Postoperative pain characteristics. | Early postoperative pain scores are recorded during postoperative hospital stay, approximately 1 year after first screening. Late ones are recorded at the one year postoperative follow-up patient contact, approximately 2 years after first screening.
  Changes from baseline in pain scores on the Visual Analog Scale at postoperative day one and two, and at 1 year postoperatively.
Duration of hospital stay after adrenalectomy. | Recorded during postoperative hospital stay, approximately 1 year after first screening.
  Number of days.
Time before return to work after adrenalectomy. | Recorded as soon as the patient goes back to work after the operation - latest at one year postoperative follow-up patient contact, approximately 2 years after first screening.
  Number of days. Applies to working study participants.
Occurrence of any surgical complications. | Early complications are recorded during postoperative hospital stay, approximately 1 year after first screening. Late ones are recorded at the one year postoperative follow-up patient contact, approximately 2 years after first screening.
  Proportion of operated patients who have had any surgical complications.
Frequency of conversion from planned laparoscopic adrenalectomy to an open procedure. | Recorded during postoperative hospital stay, approximately 1 year after first screening.
  Proportion of cases where converting to open procedure was needed.
Occurrence of any complications related to Adrenal Vein Sampling (AVS). | Early complications are recorded during and on the day after the procedure. Late ones are recorded at the one year follow-up patient contact, approximately 2 years after first screening.
  Proportion of patients who have underwent AVS and have had any complications.

CONTACTS AND LOCATIONS:
Overall Officials: Per Hellman, PhD, Principal Investigator — Uppsala University, The Department of Surgical Sciences
Locations (1):
- Uppsala University, the Department of Surgical Sciences, Uppsala, Uppsla, Sweden

IPD SHARING:
Plan to Share IPD: Undecided